CLINICAL TRIAL: NCT03503045
Title: The Rates of Overtreatment and Deintensification of Antidiabetic and Antihypertensive Medications in Patients With Diabetes Mellitus
Brief Title: The Rates of Overtreatment and Deintensification in Patients With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Prof. Dr., Gulhane School of Medicine
Other Study IDs: GSM-012018
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Polypharmacy; Overtreatment; Undertreatment
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the overtreatment and deintensification rates of antidiabetic and antihypertensive medications in patients with diabetes mellitus in Turkey.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common chronic diseases which lead to serious public health problems and a significant economic burden worldwide. The prevalence of diabetes in elderly patients is very high and is predicted to increase dramatically.

Prior studies have generally been concerned with the inadequate treatment of diabetes however, over the last few years the overtreatment of diabetes has also come to the fore. Unfortunately, there are very few data worldwide and no data in Turkey about the overtreatment of patients with type 2 diabetes.

This study aimed to assess the rates and predictors of overtreatment and undertreatment of glycemia and blood pressure in older adults with T2DM. Treatment deintensification or intensification by the physicians were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus type I or II
* Age 65 years or older
* To be under follow-up in the same center for at least one year.

Exclusion Criteria:

* Younger than 65 years old
* having decompensated liver disease
* psychiatric disorders interfering cognition or compliance
* having bariatric surgery or on renal replacement therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older and with type 1 or type 2 diabetes who were under follow-up in the same tertiary endocrine unit for at least a year were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1276 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Overtreatment for glycemia | 7 days
  HbA1c<6.5% plus use of ≥2 oral hypoglycemics or insulin, except metformine.

SECONDARY OUTCOMES:
Undertreatment for glycemia | 7 days
  HbA1c>9%
Overtreatment for blood pressure | 7 days
  systolic blood pressure < 120 mmHg or diastolic blood pressure < 65 mmHg and use of at least one drug additional to ACE inhibitors
Undertreatment for blood pressure | 7 days
  SBP≥140 mmHg or DPB ≥ 90 mmHg and use of two or less drugs
Deintensification of treatment | 7 days
  discontinuation or dosage decrease within 6 months after the index measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Sonmez, Prof.Dr., Study Director — Gulhane School of Medicine, Endocrinology and Metabolism
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No